CLINICAL TRIAL: NCT03782571
Title: Influence of Lens Design on Particulate Exchange in the Post-lens Tear Film
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6291
Record Dates: First submitted 2018-11-15; First posted 2018-12-20 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Test1/Test2/Control/Test3 (Experimental): Subjects that are adapted soft contact lens wearers between the ages of 18-40 years of age will be randomly assigned to one of four sequences. Upon completion, each subject will have worn all three lens types and been assigned the bare eye condition in both eyes.
  Interventions: Device: etafilcon a Test 1; Device: etafilcon A Test 2; Device: etafilcon A Test 3; Other: Control
- Test2/Test3/Test1/Control (Experimental): Subjects that are adapted soft contact lens wearers between the ages of 18-40 years of age will be randomly assigned to one of four sequences. Upon completion, each subject will have worn all three lens types and been assigned the bare eye condition in both eyes.
  Interventions: Device: etafilcon a Test 1; Device: etafilcon A Test 2; Device: etafilcon A Test 3; Other: Control
- Test3/Control/Test2/Test1 (Experimental): Subjects that are adapted soft contact lens wearers between the ages of 18-40 years of age will be randomly assigned to one of four sequences. Upon completion, each subject will have worn all three lens types and been assigned the bare eye condition in both eyes.
  Interventions: Device: etafilcon a Test 1; Device: etafilcon A Test 2; Device: etafilcon A Test 3; Other: Control
- Control/Test1/Test3/Test2 (Experimental): Subjects that are adapted soft contact lens wearers between the ages of 18-40 years of age will be randomly assigned to one of four sequences. Upon completion, each subject will have worn all three lens types and been assigned the bare eye condition in both eyes.
  Interventions: Device: etafilcon a Test 1; Device: etafilcon A Test 2; Device: etafilcon A Test 3; Other: Control

INTERVENTIONS:
Device: etafilcon a Test 1 — 1-DAY ACUVUE® MOIST
Device: etafilcon A Test 2 — 1-DAY ACUVUE® MOIST for ASTIGMATISM
Device: etafilcon A Test 3 — 1-DAY ACUVUE® MOIST MULTIFOCAL
Other: Control — Bare Eye

SUMMARY:
This is a 5-visit, controlled, bilateral, randomized, subject-masked, crossover (4 treatments x 4 period), non-dispensing study. Subjects will attend all study visits in their spectacle correction having not worn contact lenses on the day of the visit.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be between 18 and 40 (inclusive) years of age at the time of screening.
  4. The subject must own a wearable pair of spectacles and be willing to wear them to each study visit.
  5. The subject must be an adapted soft contact lens wearer in both eyes, having successfully worn contact lenses in the last six months by self-report.
  6. The subject must agree not to participate in other clinical research for the duration of this study.
  7. The subject's refractive cylinder must be <-1.25DC in each eye.
  8. The subject must have best corrected visual acuity of 0.20 logMAR or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or breast feeding (self-reported).
  2. Any systemic disease (e.g., Sjögren's Syndrome), infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the Investigator's discretion).
  3. Use of topical medication such as eye drops or ointment within 24 hours prior to the study visit.
  4. Any history of anaphylaxis or severe allergy.
  5. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
  6. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment
  7. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician)
  8. They have any slit lamp findings of grade 3 or higher (e.g. corneal edema, corneal neovascularization, tarsal abnormalities, conjunctival injection) or findings of < Grade 3 which in the investigator's opinion would contraindicate contact lens wear.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 subjects were enrolled into the study. Of the enrolled 9 subjects did not meet the eligibility criteria. 22 subjects completed the study and 3 subjects were discontinued from the study.
Pre-assignment Details: Subjects were randomized to 1 of 4 unique lens sequences.
Groups:
- Test 1\Control\Test 2\Test 3: Subjects randomized to this sequence received the following treatments in order: Test 1 in period 1, Control in period 2, Test 2 in period 3, and Test 3 in period 4.
- Test 2\Test 1\Test 3\Control: Subjects randomized to this sequence received the following treatments in order: Test 2 in period 1, Test 1 in period 2, Test 3 in period 3, and Control in period 4.
- Control\Test 3\Test 1\Test 2: Subjects randomized to this sequence received the following treatments in order: Control in period 1, Test 3 in period 2, Test 1 in period 3, and Test 2 in period 4.
- Test 3\Test 2\Control\Test 1: Subjects randomized to this sequence received the following treatments in order: Test 3 in period 1, Test 2 in period 2, Control in period 3, and 1 Test 1 in period 4.
Period: Period 1
Arm/Group | Test 1\Control\Test 2\Test 3 | Test 2\Test 1\Test 3\Control | Control\Test 3\Test 1\Test 2 | Test 3\Test 2\Control\Test 1
Started | 6 | 6 | 6 | 7
Completed | 5 | 6 | 6 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Test 1\Control\Test 2\Test 3 | Test 2\Test 1\Test 3\Control | Control\Test 3\Test 1\Test 2 | Test 3\Test 2\Control\Test 1
Started | 5 | 6 | 6 | 7
Completed | 5 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Test 1\Control\Test 2\Test 3 | Test 2\Test 1\Test 3\Control | Control\Test 3\Test 1\Test 2 | Test 3\Test 2\Control\Test 1
Started | 5 | 6 | 6 | 7
Completed | 3 | 6 | 6 | 7
Not Completed | 2 | 0 | 0 | 0
Not completed — Subject Unable to Attend V5 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Period 4
Arm/Group | Test 1\Control\Test 2\Test 3 | Test 2\Test 1\Test 3\Control | Control\Test 3\Test 1\Test 2 | Test 3\Test 2\Control\Test 1
Started | 3 | 6 | 6 | 7
Completed | 3 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Total: All subjects dispensed a study lens.
Arm/Group | Total
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (7.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 7
  Black or African American | 1
  White | 16
  Other | 1
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 25

OUTCOME MEASURES:

1. Primary Outcome: Microsphere Clearance Rate
Description: The rate of microsphere clearance from the post-lens tear film was assessed by the C30 image analysis metric. Where bare eye was assigned, a droplet of microsphere suspension was applied directly onto the superior temporal conjunctiva. Where lens wear was assigned, the microsphere suspension was dispensed onto the posterior concave contact lens surface immediately prior to lens application. A series of digital images were taken over a 30-minute period (every minute for the first 10 minutes and then every 5 minutes for the next 20 minutes). Data transformed from the images were calculated by the C30 image analysis metric. Higher numbers represented greater clearance. The right eye was used to evaluate microsphere clearance.
Time Frame: Post microsphere application over a 30 minute period
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol
Measure: Mean (Standard Deviation); unit: percent clearance
Units Other Than Participants: eyes
Groups:
- Test 1; Test 2; Test 3: Subjects that wore the Test 1 lens in either the first, second, third, or fourth period of the study
- Control (Bare Eye): Subjects were under the bare eye condition in either the first, second, third, or fourth period of the study.
Arm/Group | Test 1 | Test 2 | Test 3 | Control (Bare Eye)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Number analyzed (eyes) | 7 | 7 | 7 | 7
percent clearance | 96.9 (1.16) | 98.1 (2.66) | 99.4 (3.67) | 96.6 (2.68)
Statistical Analysis 1: Comparison: Test 1 vs Control (Bare Eye); Testing equivalence with respect to microsphere clearance rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; Kenward and Roger method was used for denominator degrees of freedom. Adjustment was made using a simulation-based approach; Mean Difference (Final Values) = 1.7, 99.1% CI 2-sided [-4.0 to 7.4], Standard Error of Mean 1.97 — Test 1 - Control
Statistical Analysis 2: Comparison: Test 2 vs Control (Bare Eye); Testing equivalence with respect to microsphere clearance rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.7, 99.1% CI 2-sided [-4.0 to 13.4], Standard Error of Mean 3.01 — Test 2 - Control
Statistical Analysis 3: Comparison: Test 3 vs Control (Bare Eye); Testing equivalence with respect to microsphere clearance rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.2, 99.1% CI 2-sided [-2.7 to 19.1], Standard Error of Mean 3.78 — Test 3 - Control
Statistical Analysis 4: Comparison: Test 1 vs Test 3; Testing equivalence with respect to microsphere clearance rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.5, 99.1% CI 2-sided [-2.6 to 15.5], Standard Error of Mean 3.12 — Test 3 - Test 1
Statistical Analysis 5: Comparison: Test 2 vs Test 3; Testing equivalence with respect to microsphere clearance rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.5, 99.1% CI 2-sided [-2.0 to 8.9], Standard Error of Mean 1.88 — Test 3 - Test 2
Statistical Analysis 6: Comparison: Test 1 vs Test 2; Testing equivalence with respect to microsphere clearance rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.0, 99.1% CI 2-sided [-4.3 to 10.3], Standard Error of Mean 2.54 — Test 2 - Test 1

2. Primary Outcome: Microsphere Uptake Rate
Description: The rate of microsphere uptake into the post-lens tear film was assessed by the U5 image analysis metric. Where bare eye was assigned, a droplet of microsphere suspension was applied directly onto the superior temporal conjunctiva. Where a lens was assigned the lens was applied and after a 10-minute settling period, a droplet of microsphere suspension was applied directly to the superior temporal conjunctiva. A series of digital images were taken over a 10-minute period (every minute for 10 minutes). Data transformed from the images were calculated by the U5 image analysis metric. Higher numbers represented greater uptake rate. The left eye was used to evaluate microsphere uptake.
Time Frame: Post microsphere application over a 10 minute period
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol
Measure: Mean (Standard Deviation); unit: percent uptake
Units Other Than Participants: eyes
Arm/Group | Test 1 | Test 2 | Test 3 | Control (Bare Eye)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Number analyzed (eyes) | 7 | 7 | 7 | 7
percent uptake | 8.5 (4.09) | 6.8 (5.31) | 2.9 (3.35) | 1.5 (7.62)
Statistical Analysis 1: Comparison: Test 1 vs Control (Bare Eye); Testing equivalence with respect to microsphere uptake rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.4, 99.1% CI 2-sided [-1.0 to 17.8], Standard Error of Mean 3.24 — Test 1 - Control
Statistical Analysis 2: Comparison: Test 2 vs Control (Bare Eye); Testing equivalence with respect to microsphere uptake rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.6, 99.1% CI 2-sided [-7.8 to 20.9], Standard Error of Mean 4.95 — Test 2 - Control
Statistical Analysis 3: Comparison: Test 3 vs Control (Bare Eye); Testing equivalence with respect to microsphere uptake rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.9, 99.1% CI 2-sided [-15.1 to 20.9], Standard Error of Mean 6.22 — Test 3 - Control
Statistical Analysis 4: Comparison: Test 1 vs Test 3; Testing equivalence with respect to microsphere uptake rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.5, 99.1% CI 2-sided [-20.4 to 9.4], Standard Error of Mean 5.13 — Test 3 - Test 1
Statistical Analysis 5: Comparison: Test 2 vs Test 3; Testing equivalence with respect to microsphere uptake rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.7, 99.1% CI 2-sided [-12.6 to 5.3], Standard Error of Mean 3.10 — Test 3 - Test 2
Statistical Analysis 6: Comparison: Test 1 vs Test 2; Testing equivalence with respect to microsphere uptake rate; Test type: Equivalence — Equivalence is concluded if the upper limit is less than 10% and the lower limit is greater than -10%; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.8, 99.1% CI 2-sided [-13.9 to 10.3], Standard Error of Mean 4.18 — Test 2 - Test 1

3. Secondary Outcome: Lens Movement
Description: Lens movement was assessed for primary gaze, up-gaze, and push up by clinical grading. Primary gaze movement was evaluated by observing the vertical movement of the contact lens that occurs with a full blink without manipulating the subject's lids. Up-gaze movement was assessed by estimating the vertical lens movement observed when the subject looks up and blinks fully without manipulating the subject's lids. The push-up test consists of a gentle digital push of the lens upwards using the lower lid. The resistance of the lens to of the lens to upward movement is judged. Lens movement was graded according to the following scale: Excessive (+2), Moderate movement (+1), Optimal (0), Minimal (-1), and Insufficient (-2). All available data for lens movement in the safety population were reported.
Time Frame: Post microsphere application at 30-minute timepoint (OD); post microsphere application at 10-minute timepoint (OS)
Population: All subjects dispensed a study lens.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Test 1 | Test 2 | Test 3
Number analyzed (Participants) | 25 | 24 | 22
Number analyzed (eyes) | 47 | 44 | 43
eyes
  Primary Position: Insufficient(-2) | 0 | 1 | 2
  Primary Position: Minimal(-1) | 12 | 7 | 10
  Primary Position: Optimal(0) | 28 | 27 | 24
  Primary Position: Moderate(+1) | 7 | 9 | 7
  Primary Position: Excessive(+2) | 0 | 0 | 0
  Push Up: Insufficient(-2) | 0 | 1 | 1
  Push Up: Minimal(-1) | 6 | 6 | 2
  Push Up: Optimal(0) | 31 | 30 | 28
  Push Up: Moderate(+1) | 10 | 7 | 12
  Push Up: Excessive(+2) | 0 | 0 | 0
  Up-gaze: Insufficient(-2) | 0 | 1 | 2
  Up-gaze: Minimal(-1) | 18 | 12 | 9
  Up-gaze: Optimal(0) | 22 | 20 | 24
  Up-gaze: Moderate(+1) | 7 | 11 | 8
  Up-gaze: Excessive(+2) | 0 | 0 | 0

4. Secondary Outcome: Corneal Curvature
Description: Corneal curvature was assessed by Visante™ OCT. The following were measured: Sclera Angle-Temporal and Sclera Angle-Nasal.
Time Frame: Baseline
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: Degree
Units Other Than Participants: eyes
Arm/Group | Total
Number analyzed (Participants) | 25
Number analyzed (eyes) | 50
Degree
  Sclera Angle-Temporal | 39.14 (2.374)
  Sclera Angle-Nasal | 36.64 (3.311)

5. Secondary Outcome: Corneal Curvature
Description: Corneal curvature was assessed by Visante™ OCT. Sagital Height was measured.
Time Frame: Baseline
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: eyes
Arm/Group | Total
Number analyzed (Participants) | 25
Number analyzed (eyes) | 50
Millimeter | 3.700 (0.1854)

6. Secondary Outcome: Blink Rate
Description: Blinking characteristics were captured using an infra-red camera (FLIR Grasshopper 3 camera) and infra-red LED illumination (Thorlabs LIU780A). During video capture the subject was directed to view a wildlife video on an Ipad at a working distance of approximately 1 meter. The infrared video was captured for 3 minutes at 500 frames per second. Subsequent video analysis recorded the blink rate (blinks per minute) over the 3-minute period. Baseline values were reported across all subjects who were dispensed a study lens. Blink rate post microsphere application was reported by treatment. All available data for blink rate in the safety population were reported.
Time Frame: Baseline and the 30-minute post microsphere application time point in the right eye and at the 10-minute post microsphere application timepoint in the left eye.
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: blinks per minute
Units Other Than Participants: eyes
Arm/Group | Test 1 | Test 2 | Test 3 | Control (Bare Eye) | Total
Number analyzed (Participants) | 25 | 24 | 22 | 24 | 25
Number analyzed (eyes) | 47 | 44 | 42 | 48 | 50
blinks per minute
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 28.2 (16.48)
  Post Lens Insertion | 23.3 (11.63) | 26.1 (15.88) | 25.0 (13.02) | 19.8 (13.08) | 0 (0)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 13 weeks.
Groups:
- Control (Bare Eye): Subjects were under bare eye condition in either the first, second, third, or fourth period of the study.
Arm/Group | Test 1 | Test 2 | Test 3 | Control (Bare Eye)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1 (N=25) | Test 2 (N=25) | Test 3 (N=25) | Control (Bare Eye) (N=25)
Unconfirmed Corneal Endothelium Keratic Precipitate (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unconfirmed Corneal Endothelium Keratic Precipitate was reported in the right eye. The adverse event was deemed unrelated to the study by the investigator and the subject was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03782571/Prot_SAP_000.pdf